CLINICAL TRIAL: NCT04658342
Title: Effects of Oral Cancer Treatments on Upper Esophageal Opening During Swallowing
Status: Terminated | Type: Observational
Why Stopped: per Slow Accrual
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0495; SMPH/SURGERY/OTOLARYNGOLOGY (Other: UW Madison); A539770 (Other: UW Madison); Protocol Version 4/26/2022 (Other: UW Madison); UW20051 (Other: UWCCC)
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Cancer of Head and Neck
Keywords: quality of life; swallowing outcomes; oral cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Mouth Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oral Cancer Patients
  Interventions: Diagnostic Test: Videofluoroscopic imaging (VFSS) with high-resolution manometry (HRM)

INTERVENTIONS:
Diagnostic Test: Videofluoroscopic imaging (VFSS) with high-resolution manometry (HRM) — The Videofluoroscopic Imaging (VFSS) is done by inserting a small catheter into the nose and down the throat. The catheter is approximately .4 millimeters in diameter. A trained speech-language pathologist will insert the catheter after applying numbing medicine, or topical anesthetic, inside the nose.
  The high-resolution manometry (HRM) is a swallowing pressure test done at the same time as the VFSS. The HRM will measure how strong the throat muscle squeeze the liquids and foods that a person swallows.
  The VFSS and HRM will occur about one month after surgery and three months after the completion of the radiation treatment.

SUMMARY:
The purpose of this study is to investigate post-operative and post-radiation upper esophageal sphincter opening measures in oral cancer patients, compare measures to age- and gender-matched healthy adults, and determine relationships with patient swallowing outcomes and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Oral cancer that includes tongue or floor of mouth clinical stage T1 or higher
* May have disease that extends to base of tongue or other site as long as floor of mouth or tongue are involved
* Adults at least 18 years of age

Exclusion Criteria:

* Oral cancer of the lip, cheek, palate or other site not impacting tongue or floor of mouth musculature
* History of floor of mouth, tongue base, pharyngeal or laryngeal surgical resection
* History of radiation treatment to the head and neck
* History of dysphagia prior to onset of oral cancer symptoms
* Allergy to lidocaine, barium, adhesive tape or apple flavoring
* Woman of childbearing years who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population are patients with a diagnosis of oral and neck cancer that are selected at the primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-03-25 (Actual)

PRIMARY OUTCOMES:
Change in Upper Esophageal Maximum Admittance as measured by HRM among time points of oral cancer treatment. | Approximately 4 weeks (post-surgery), and up to 6 months (3 months post-radiation)
  This measure provides understanding of how well throat muscles pull the upper esophagus open to allow flow of liquid or food from the throat to the esophagus.
Change in Upper Esophageal Integrated Relaxation Pressure (IRP) as measured by HRM | Approximately 4 weeks (post-surgery), and up to 6 months (3 months post-radiation)
  This measure indicates how well the muscles of the upper esophageal sphincter relax to allow liquid and food to pass through.
Change in Hypopharyngeal Pressure at Nadir Impedence (PNI) as measured by HRM | Approximately 4 weeks (post-surgery), and up to 6 months (3 months post-radiation)
  This measure indicates how well the upper esophagus stretches open to accept the liquid or food.

SECONDARY OUTCOMES:
Change in the MD Anderson Dysphagia Inventory (MDADI) Scores among time points of oral cancer treatment | Approximately 4 weeks (post-surgery), and up to 6 months (3 months post-radiation)
  Measurement of swallowing-related quality of life. This patient-rated tool has a maximum score of 100 points total across 20 questions, where the highest score indicates better overall swallow-related quality of life.
Dynamic Imaging Grade of Swallowing Toxicity (DIGEST) Grading Scale Score | Approximately 4 weeks (post-surgery), and up to 6 months (3 months post-radiation)
  Dynamic Imaging Grade of Swallowing Toxicity (DIGEST) grade of 0 to 4, where lower grade reflects better swallow function
Statistical Correlation between MDADI and Maximum Admittance | Approximately 4 weeks (post-surgery), and up to 6 months (3 months post-radiation)
Statistical Correlation between DIGEST and Maximun Admittance | Approximately 4 weeks (post-surgery), and up to 6 months (3 months post-radiation)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Thibeault, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No